CLINICAL TRIAL: NCT02908529
Title: Effect of Atomoxetine and Oxybutynin on Phenotype Traits and OSA Severity
Brief Title: Atomoxetine and Oxybutynin in Obstructive Sleep Apnea
Acronym: ATOSA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Assistant Professor of Medicine - Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BWH-2014P001033
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — oxybutynin; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 2 hours before bedtime
  Interventions: Drug: Placebo, 2 tablets
- Combination product of Atomoxetine and Oxybutynin (Active Comparator): Combination product of Atomoxetine 80 mg and Oxybutynin 5 mg 2 hours before sleep
  Interventions: Drug: Combination product of Atomoxetine and Oxybutynin

INTERVENTIONS:
Drug: Combination product of Atomoxetine and Oxybutynin — Combination product of Atomoxetine 80 mg and Oxybutynin 5 mg 2 hours before sleep
  Other Names: Strattera + Ditropan
  Arms: Combination product of Atomoxetine and Oxybutynin
Drug: Placebo, 2 tablets — Placebo 2 tablets 2 hours before sleep
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal subjects. Until recently, the search for medicines to activate pharyngeal muscles in sleeping humans has been discouraging. However, exciting new animal research has shown that drugs with noradrenergic and antimuscarinic effects can restore pharyngeal muscle activity to waking levels. In this protocol the investigators will test the effect of atomoxetine (a norepinephrine reuptake inhibitor) and oxybutynin (an antimuscarinic drug) administered together on OSA phenotype traits and OSA severity during sleep.

ELIGIBILITY:
Inclusion Criterion:

- AHI > 20

Exclusion Criteria:

* Any medical condition other than well controlled hypertension.
* Any medication known to influence breathing, sleep/arousal or muscle physiology.
* Claustrophobia.
* Inability to sleep supine.
* Allergy to lidocaine, Oxymetazoline HCl, atomoxetine/oxybutynin.
* Individuals with underlying cardiac disease, such as arrhythmias.
* Individuals taking psychiatric medications, such as atomoxetine, or any of the studied medications for medical care.
* History of seizures
* For women: Pregnancy.
* History of panic disorder / hyperventilation syndrome / Attention deficit-hyperactivity disorder (ADHD) / autism

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Taranto-Montemurro L, Messineo L, Sands SA, Azarbarzin A, Marques M, Edwards BA, Eckert DJ, White DP, Wellman A. The Combination of Atomoxetine and Oxybutynin Greatly Reduces Obstructive Sleep Apnea Severity. A Randomized, Placebo-controlled, Double-Blind Crossover Trial. Am J Respir Crit Care Med. 2019 May 15;199(10):1267-1276. doi: 10.1164/rccm.201808-1493OC. PMID 30395486

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Ato-Oxy Second: Placebo-matching ato-oxy administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then ato-oxy administered 30 mins before normal sleep time on second study night.
- Ato-Oxy First, Placebo Second: Ato-Oxy administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then placebo administered 30 mins before normal sleep time on second study night.
Period: Overall Study
Arm/Group | Placebo First, Ato-Oxy Second | Ato-Oxy First, Placebo Second
Started | 10 | 12
Completed | 10 | 10
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized, completed both study nights, and were included in the analysis.
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [46 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI, Events/Hour of Sleep)
Description: Based on previous studies the investigators anticipate that Atomoxetine and Oxybutynin will reduce AHI more effectively in subjects with moderate sleep apnea, mildly obese (BMI<32), Vpassive > 50% of Veupnea (ventilation during eupneic ventilatory drive), low muscle compensation (Vactive - Vpassive <1 L/min)
Time Frame: 1 night
Population: 2 participants were not analyzed because they dropped out between the 2 intervention arms
Measure: Median (Inter-Quartile Range); unit: events/hours of sleep
Groups:
- Placebo: Placebo (2 tablets) 30 minutes hours before bedtime
- Combination Product of Atomoxetine and Oxybutynin: Combination product of Atomoxetine 80 mg and Oxybutynin 5 mg 30 minutes before sleep
Arm/Group | Placebo | Combination Product of Atomoxetine and Oxybutynin
Number analyzed (Participants) | 20 | 20
events/hours of sleep | 28.5 [10.9 to 51.6] | 7.5 [2.4 to 18.6]
Statistical Analysis 1: Comparison: Placebo vs Combination Product of Atomoxetine and Oxybutynin; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -15.9

2. Secondary Outcome: Genioglossus Muscle Responsiveness to Increased Ventilatory Drive (Esophageal Pressure Swings)
Description: For genioglossus muscle responsiveness, data will be expressed as change in electromyography of genioglossus (GG EMG) for cmH2O change in esophageal pressure.
Time Frame: 1 night
Population: 4 patients did not accept to perform intramuscular EMG measurement (genioglossus electromyography) 2 patients were not analyzed because they dropped out after the first arm of the study
Measure: Median (Inter-Quartile Range); unit: %GG/cmH2O
Arm/Group | Placebo | Combination Product of Atomoxetine and Oxybutynin
Number analyzed (Participants) | 16 | 16
%GG/cmH2O | 2.2 [1.1 to 4.7] | 6.3 [3.0 to 18.3]

ADVERSE EVENTS:
Time Frame: 1 night
Description: All randomized participants who received at least one dose of desipramine or placebo.
Groups:
- Placebo: Placebo 2 capsules 30 mins before bedtime
- Combination Product of Atomoxetine and Oxybutynin: Combination product of Atomoxetine 80 mg and Oxybutynin 5 mg 30 mins before sleep
Arm/Group | Placebo | Combination Product of Atomoxetine and Oxybutynin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Combination Product of Atomoxetine and Oxybutynin (N=20)
delayed micturition (Renal and urinary disorders) | 0 (0) | 2 (2)
Dry mouth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
insomnia (Nervous system disorders) | 3 (3) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT02908529/Prot_SAP_000.pdf